CLINICAL TRIAL: NCT01349049
Title: A Phase 1/2 Safety and Efficacy Study of Orally Administered PLX3397 in Adults With Relapsed or Refractory FLT3-ITD Positive Acute Myeloid Leukemia (AML)
Brief Title: Phase 1/2 Safety and Efficacy of PLX3397 in Adults With Relapsed or Refractory Acute Myeloid Leukemia (AML)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: Plexxikon (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PLX108-05
Record Dates: First submitted 2011-05-04; First posted 2011-05-06 (Estimated); Results first posted 2019-11-21 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML; relapsed; refractory
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence | interventions — pexidartinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (9):
- oral dose of 3000 mg/day PLX3397 (RP2D) (Experimental): Subjects will be dosed at the recommended Phase 2 dose (RP2D)
  Interventions: Drug: PLX3397
- oral dose of 800 mg/day of PLX3397 (Experimental): Level 0
  Interventions: Drug: PLX3397
- oral dose of 1000 mg/day PLX3397 (Experimental): Level 1
  Interventions: Drug: PLX3397
- oral dose of 1200 mg/day PLX3397 (Experimental): Level 2
  Interventions: Drug: PLX3397
- oral dose of 1400 mg/day PLX3397 (Experimental): Level 3
  Interventions: Drug: PLX3397
- oral dose of 2000 mg/day PLX3397 (Experimental): Level 4
  Interventions: Drug: PLX3397
- oral dose of 3000 mg/day PLX3397 (Experimental): Level 5
  Interventions: Drug: PLX3397
- oral dose of 4000 mg/day PLX3397 (Experimental): Level 6
  Interventions: Drug: PLX3397
- oral dose of 5000 mg/day PLX3397 (Experimental): Level 7
  Interventions: Drug: PLX3397

INTERVENTIONS:
Drug: PLX3397 — Maximum Tolerated Dose of PLX3397 will be administered orally, twice daily.
  Other Names: Plexxikon 3397
  Arms: oral dose of 3000 mg/day PLX3397 (RP2D)
Drug: PLX3397 — The drug product is available in capsule form, to be taken orally.
  Other Names: Plexxikon 3397
  Arms: oral dose of 1000 mg/day PLX3397; oral dose of 1200 mg/day PLX3397; oral dose of 1400 mg/day PLX3397; oral dose of 2000 mg/day PLX3397; oral dose of 3000 mg/day PLX3397; oral dose of 4000 mg/day PLX3397; oral dose of 5000 mg/day PLX3397; oral dose of 800 mg/day of PLX3397

SUMMARY:
The purpose of this study is to evaluate the safety of study drug PLX3397 at 3 dose levels (800 mg/day, 1000 mg/day, and 1200 mg/day) and explore the efficacy in patients with relapsed or refractory acute myeloid leukemia (AML). Additional dose levels beyond 1200 mg/day may be considered based on safety and efficacy observations.

DETAILED DESCRIPTION:
Protocol PLX108-05 is a Phase 1/2 open-label, sequential dose escalation (Part 1) followed by cohort expansion (Part 2) design at the recommended phase 2 dose established in Part 1 (i.e. 3,000 mg/day). Treatment with PLX3397 will consist of continuous oral administration in 28-day cycles until unacceptable or dose-limiting toxicity, disease progression or relapse, patient death, Investigator decision, or voluntary withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥18 years old.
* Morphologically documented primary Acute Myeloid Leukemia (AML), prior-chemotherapy-related AML or AML secondary to an antecedent hematologic disorder (e.g., Myelodysplastic Syndrome) as defined by World Health Organization criteria, confirmed by pathology review. For Cohort Expansion Phase (Part 2) only: Bone marrow involvement is required.
* Have either relapsed or refractory AML, or who have newly diagnosed Flt3-ITD positive AML but either refuse or are considered by the Investigator not to be an appropriate candidate for standard chemotherapy.

  1. Relapsed disease is defined as the reappearance of leukemia cells in the bone marrow or peripheral blood or elsewhere in the body (other tissues/organs) after the attainment of a CR.
  2. Refractory disease is defined by the failure to obtain a complete remission (CR) with a High-Dose Cytarabine (HDAC)-containing or a standard induction regimen. Patients who require two cycles of induction therapy to attain a first CR are not considered to have refractory disease.
* Positive for Flt3-ITD activating mutations during Screening. Local laboratory results must be received prior to enrollment. Patients with a history of Flt3-ITD positive disease may be considered after discussion with the Medical Monitor.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
* Adequate recovery (to at least Grade 1) from toxicity of prior therapy as follows:

  1. ≥2 weeks for cytotoxic therapy (except hydroxyurea, which is permitted at doses of ≤5g/day during the first 2 weeks of Cycle 1) prior to C1D1.
  2. ≥4 half-lives for non-cytotoxic therapy prior to C1D1. Patients must have a wash-out period from their last chemotherapy of either ≥2 weeks OR at least 4 half-lives prior to C1D1. For patients whose most recent anti-tumor treatment regimen consisted of a multi-agent cocktail, the patient must have a wash-out period of at least 4 half-lives of the agent with the longest half-life.
* Adequate hepatic and renal function

  1. Adequate renal function, defined as Creatinine Clearance >60 mL/min or serum creatinine of ≤ 1.3 mg/dL (115 μM).
  2. Adequate hepatic function, defined as Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤3.0X Upper limit of normal (ULN) and serum direct bilirubin ≤1.5X ULN. Exceptions may be made for patients with elevated liver transaminases secondary to AML after discussion with the Medical Monitor
* Life expectancy of at least 1 month
* Willing and able to provide written informed consent prior to any study related procedures and to comply with all study requirements and for 3 months after last dose.
* Women of child-bearing potential must have a negative pregnancy test within 7 days of initiation of dosing and must agree to use two acceptable methods of birth control while on study drug and for 3 months after the last dose. Women of non-childbearing potential may be included if they meet at least one of the following criteria:

  1. Surgically sterile
  2. Have been postmenopausal for ≥1 year
  3. Have Follicle Stimulating Hormone (FSH) levels indicative of postmenopausal state (i.e., 30-120 IU/L) documented within 21 days of C1D1.

Sexually active men must also agree to use an acceptable method of birth control while on study drug and for at least 3 months after the last dose

Exclusion Criteria:

* Diagnosis of acute promyelocytic leukemia
* Diagnosis of chronic myelogenous leukemia in blast crisis
* Presence of central nervous system (CNS) involvement of leukemia. Patients with a history of CNS involvement may be considered after discussion with the Medical Monitor
* Patients eligible for Hematopoietic Stem Cell Transplantation (HSCT) at the time of screening. However, patients who meet one or both of the following criteria may be eligible for study participation:

  1. Patients who are eligible for HSCT but with non-optimal AML disease control (i.e., blasts > 5%) may be enrolled into this study as a bridge-to-transplant.
  2. Patients with relapsed disease following a prior HSCT may be enrolled into this study as an alternative to a second HSCT or as a bridge-to-transplant regimen.
* For both Parts 1 and 2, receipt of HSCT within 60 days of the first dose of PLX3397 is an exclusion criterion. Patients on immunosuppressive therapy post HSCT, or with clinically significant graft-versus-host disease are excluded from Part 1. (Use of topical steroids for ongoing skin Graft vs. host disease [GVHD] is permitted). Patients for Part 1 must have a wash-out period of ≥2 weeks or at least 4 half-lives from their last systemic immunosuppressive treatment for Graft vs. host disease. Patients for Part 2 may be receiving systemic immunosuppressive treatment for management of GVHD at the time of screening and enrollment
* Investigational drug use within 28 days of the first dose of PLX3397
* For Cohort Expansion Phase (Part 2) only: Patients who are positive for the D835 mutation at Screening are excluded.
* A concurrent active cancer that requires non-surgical therapy (e.g., chemotherapy, radiation, adjuvant therapy). Prior history of other cancer is allowed, as long as there is no active disease within 1 year of the first dose of PLX3397.
* Refractory nausea and vomiting, malabsorption, biliary shunt significant bowel resection, GVHD affecting the gut, or any other condition that would preclude adequate absorption
* Patients with serious illnesses, uncontrolled infection, medical conditions, or other medical history including abnormal laboratory results, which in the investigator's opinion would be likely to interfere with a patient's participation in the study, or with the interpretation of the results
* Women of child-bearing potential who are pregnant or breast feeding
* At Screening, QT interval, Frederica's formula (QTcF) >450 msec for males; QTcF >470 msec for females
* Patients with a history of D835 mutations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2011-11-21 (Actual); Primary Completion 2015-01-20 (Actual); Study Completion 2018-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Olga Frankfurt, MD, Principal Investigator — Robert H. Lurie Comprehensive Cancer Center of Northwestern University - Chicago, IL; Mark Levis, MD, PhD, Principal Investigator — Johns Hopkins University; John Pagel, MD, PhD, Principal Investigator — Fred Hutchinson Cancer Research Center - Seattle, WA; Alexander Perl, MD, Principal Investigator — Hospital of the University of Pennsylvania - Philadelphia, PA; Gail Roboz, MD, Principal Investigator — Weill Cornell Medical College/New York Presbyterian Hospital - New York, NY; Catherine Smith, MD, Principal Investigator — University of California Medical Center - San Francisco, CA; Richard Stone, MD, Principal Investigator — Dana-Farber Cancer Institute - Boston, MA; Eunice Wang, MD, Principal Investigator — Roswell Park Cancer Institute - Buffalo, NY
Locations (9):
- United States (9):
  - UCSF Helen Diller Family Family Comprehensive Cancer Center, San Francisco, California
  - Northwestern University, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - New York Presby Hospital, Weill Medical College at Cornell University, New York, New York
  - University of Pennsylvania, Abramson Cancer Center, Philadelphia, Pennsylvania
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Smith CC, Levis MJ, Frankfurt O, Pagel JM, Roboz GJ, Stone RM, Wang ES, Severson PL, West BL, Le MH, Kayser S, Lam B, Hsu HH, Zhang C, Bollag G, Perl AE. A phase 1/2 study of the oral FLT3 inhibitor pexidartinib in relapsed/refractory FLT3-ITD-mutant acute myeloid leukemia. Blood Adv. 2020 Apr 28;4(8):1711-1721. doi: 10.1182/bloodadvances.2020001449. PMID 32330242

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 90 participants (34 in Part 1 and 56 in part 2) were enrolled in the study and received PLX3397.
Pre-assignment Details: The study participants enrolled are patients with relapsed or refractory Flt3-ITD+ AML, or newly diagnosed Flt3-ITD + AML patients who either refused or were considered not to be appropriate candidates for chemotherapy.
Groups:
- Part 1: 800 mg/Day: Participants with acute myeloid leukemia (AML), either relapsed/refractory or newly diagnosed and unfit to receive chemotherapy, received PLX3397 800 mg/day
- Part 1: 1000 mg/Day: Participants with acute myeloid leukemia (AML), either relapsed/refractory or newly diagnosed and unfit to receive chemotherapy, received PLX3397 1000 mg/day
- Part 1: 1200 mg/Day: Participants with acute myeloid leukemia (AML), either relapsed/refractory or newly diagnosed and unfit to receive chemotherapy, received PLX3397 1200 mg/day
- Part 1: 1400 mg/Day: Participants with acute myeloid leukemia (AML), either relapsed/refractory or newly diagnosed and unfit to receive chemotherapy, received PLX3397 1400 mg/day.
- Part 1: 2000 mg/Day: Participants with acute myeloid leukemia (AML), either relapsed/refractory or newly diagnosed and unfit to receive chemotherapy, received PLX3397 2000 mg/day.
- Part 1: 3000 mg/Day; Part 2: 3000 mg/Day: Participants with acute myeloid leukemia (AML), either relapsed/refractory or newly diagnosed and unfit to receive chemotherapy, received PLX3397 3000 mg/day.
- Part 1: 4000 mg/Day: Participants with acute myeloid leukemia (AML), either relapsed/refractory or newly diagnosed and unfit to receive chemotherapy, received PLX3397 4000 mg/day.
- Part 1: 5000 mg/Day: Participants with acute myeloid leukemia (AML), either relapsed/refractory or newly diagnosed and unfit to receive chemotherapy, received PLX3397 5000 mg/day.
Period: Overall Study
Arm/Group | Part 1: 800 mg/Day | Part 1: 1000 mg/Day | Part 1: 1200 mg/Day | Part 1: 1400 mg/Day | Part 1: 2000 mg/Day | Part 1: 3000 mg/Day | Part 1: 4000 mg/Day | Part 1: 5000 mg/Day | Part 2: 3000 mg/Day
Started | 3 | 7 | 3 | 3 | 3 | 6 | 5 | 4 | 56
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not Completed | 3 | 7 | 3 | 3 | 3 | 6 | 5 | 4 | 55
Not completed — Disease progression | 3 | 5 | 3 | 2 | 2 | 2 | 3 | 2 | 33
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 3 | 1 | 0 | 4
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Hematopoietic stem cell transplant | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 4
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 5
Not completed — Non-compliance | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: 800 mg/Day | Part 1: 1000 mg/Day | Part 1: 1200 mg/Day | Part 1: 1400 mg/Day | Part 1: 2000 mg/Day | Part 1: 3000 mg/Day | Part 1: 4000 mg/Day | Part 1: 5000 mg/Day | Part 2: 3000 mg/Day | Total
Number analyzed (Participants) | 3 | 7 | 3 | 3 | 3 | 6 | 5 | 4 | 56 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.0 (28.2) | 56.7 (18.5) | 65.7 (12.9) | 61.7 (19.7) | 70.7 (11.2) | 61.0 (9.7) | 54.8 (14.5) | 63.8 (2.5) | 55.9 (14.6) | 57.7 (14.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 5 | 2 | 2 | 1 | 4 | 4 | 3 | 23 | 44
  Male | 3 | 2 | 1 | 1 | 2 | 2 | 1 | 1 | 33 | 46
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 4 | 1 | 0 | 0 | 1 | 1 | 0 | 7 | 14
  White | 2 | 2 | 2 | 2 | 3 | 5 | 3 | 2 | 35 | 56
  More than one race | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 11 | 15
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 7 | 3 | 3 | 3 | 6 | 5 | 4 | 56 | 90

OUTCOME MEASURES:

1. Primary Outcome: Summary of Best Modified Criteria Response Results, Bridged-to-Transplant (BTT) Participants, and Composite Remission Rates in Patients on Treatment With PLX3397 (Dose Expansion, Part 2).
Description: Complete remission (CR): Has bone marrow regenerating normal cells, achieve a morphologic leukemia-free state, Complete remission with incomplete platelet recovery (CRp): CR except for incomplete platelet recovery, Complete remission with incomplete recovery (CRi): CR except for incomplete hematological recovery with residual neutropenia, Partial response (PR): bone marrow generates normal hematopoietic cells, evidence of peripheral recovery with no or a few regenerating circulating blasts. Decrease of ≥50% of blasts in bone marrow aspirate, total marrow blasts between 5% -25%, Non-response (NR) were assessed using modified International Working Group (IWG) response criteria for AML. Successfully (BTT) patients and successfully BTT patients (CR, CRp, or CRi) are also reported. Successfully BTT is defined as any patient who discontinued PLX3397 treatment specifically for the purpose of undergoing a hematopoietic stem cell transplant and who subsequently received the planned transplant.
Time Frame: 1 year post dose
Population: Efficacy analyses were conducted in the Part 2 Efficacy Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: 3000 mg/Day
Number analyzed (Participants) | 56
Participants
  CR | 1
  CRp | 1
  CRi | 4
  PR | 5
  NR | 45
  Successful BTT patients | 4
  Successful BTT patient (CR, CRp, or CRi) | 8

2. Primary Outcome: Summary of Time-to-Event Endpoints in Patients on Treatment With PLX3397 (Dose Expansion, Part 2)
Description: Median survival estimates were based on the Kaplan-Meier method. In the event disease progression/relapse or death was not documented prior to study termination, endpoints were censored at the date of last evaluable tumor assessment. Duration of remission, duration of complete remission, and disease-free survival, initial response was based on the modified response criteria. Duration of complete remission was defined as the number of days from the date of initial CR, CRp, or CRi response to the date of first documented disease relapse or death, whichever occurred first. Disease-free survival was defined as the number of days from the date of initial CR, CRp, or CRi to the date of documented disease relapse or death from any cause, whichever occurred first.
Time Frame: 1 year post dose
Population: Time-to-event analyses were assessed in the Part 2 Efficacy Population.
Measure: Median (90% Confidence Interval); unit: days
Arm/Group | Part 2: 3000 mg/Day
Number analyzed (Participants) | 56
days
  Duration of remission | 91 [43 to 337]
  Duration of complete remission | 289 [289 to 289]
  Progression-free survival | 48 [30 to 58]
  Disease-free survival | 289 [289 to 289]
  Overall survival | 112 [77 to 150]

3. Secondary Outcome: Number of Participants With On-treatment Best Modified Criteria Response Results of Partial Remission (PR) During Treatment With PLX3397 (Dose Expansion, Part 2)
Description: Modified International Working Group Response Criteria for Acute Myeloid Leukemia defines Partial Remission (PR) as the following: Partial Remission (PR): Patients must have bone marrow regenerating normal hematopoietic cells with evidence of peripheral recovery with no (or only a few regenerating) circulating blasts and with a decrease of at least 50% in the percentage of blasts in the bone marrow aspirate with the total marrow blasts between 5% and 25%. In addition, patients do not need to be Red Blood Cell (RBC) or platelet transfusion independent.
Time Frame: 1 year post dose
Population: Efficacy analyses were conducted in the Part 2 Efficacy Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: 3000 mg/Day
Number analyzed (Participants) | 56
Participants | 5

4. Secondary Outcome: Number of Participants With On-treatment Best Classic Criteria Response Results During Treatment With PLX3397 (Dose Expansion, Part 2)
Description: Complete Remission (CR):
  Bone marrow blasts <5%; absence of blasts with Auer rods; absence of extramedullary disease; absolute neutrophil count >1.0 x 109/L (1000/μL); platelet count >100 x 109/L (100000/μL); red cell transfusion independent
  CR with incomplete recovery (CRi):
  All CR criteria except for residual neutropenia (<1.0 x 109/L) or thrombocytopenia
  Partial Remission (PR):
  All hematologic criteria of CR; decrease of bone marrow blast percentage to 5-25%; decrease of pretreatment bone marrow blast percentage by at least 50%.
Time Frame: 1 year post dose
Population: Efficacy analyses were conducted in the Part 2 Efficacy Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: 3000 mg/Day
Number analyzed (Participants) | 56
Participants
  CR | 2
  CRi | 6
  PR | 2
  NR | 46

5. Secondary Outcome: Number of Participants Reporting an Incidence of Adverse Events During Treatment With PLX3397 (Part 1, Dose Escalation and Part 2, Dose Expansion)
Time Frame: 1 year post dose
Population: Adverse events were assessed in the Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: 800 mg/Day | Part 1: 1000 mg/Day | Part 1: 1200 mg/Day | Part 1: 1400 mg/Day | Part 1: 2000 mg/Day | Part 1: 3000 mg/Day | Part 1: 4000 mg/Day | Part 1: 5000 mg/Day | Part 2: 3000 mg/Day
Number analyzed (Participants) | 3 | 7 | 3 | 3 | 3 | 6 | 5 | 4 | 56
Participants
  At least 1 AE | 3 | 7 | 3 | 3 | 3 | 6 | 5 | 4 | 56
  At least 1 treatment-related AE | 2 | 4 | 3 | 3 | 3 | 4 | 4 | 4 | 49
  AE that lead to change in drug administration | 0 | 4 | 2 | 1 | 2 | 5 | 4 | 3 | 28
  At least 1 AE with CTCAE Grade >=3 | 3 | 7 | 2 | 3 | 2 | 5 | 5 | 4 | 50
  Serious Adverse Event (SAE)or other significant AE | 1 | 5 | 2 | 1 | 2 | 5 | 4 | 4 | 39
  At least 1 treatment-related Serious Adverse Event | 0 | 2 | 0 | 1 | 1 | 1 | 0 | 1 | 10
  AE resulting in death | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 9
  SAE leading to discontinuation of study drug | 0 | 2 | 0 | 0 | 0 | 3 | 2 | 0 | 9

6. Secondary Outcome: Number of Participants Reporting an Incidence of Treatment-Related Treatment Emergent Adverse Events During Treatment With PLX3397 (Dose Escalation, Part 1 and Dose Expansion, Part 2)
Description: Data reported are Treatment-Related Treatment Emergent Adverse Events that are ≥15% Occurrence in all patients.
Time Frame: 1 year post dose
Population: Adverse events were assessed in the Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: 800 mg/Day | Part 1: 1000 mg/Day | Part 1: 1200 mg/Day | Part 1: 1400 mg/Day | Part 1: 2000 mg/Day | Part 1: 3000 mg/Day | Part 1: 4000 mg/Day | Part 1: 5000 mg/Day | Part 2: 3000 mg/Day
Number analyzed (Participants) | 3 | 7 | 3 | 3 | 3 | 6 | 5 | 4 | 56
Participants
  At least 1 treatment-related AE | 2 | 4 | 3 | 3 | 3 | 4 | 4 | 4 | 49
  Nausea | 2 | 1 | 2 | 3 | 0 | 2 | 1 | 3 | 21
  Diarrhoea | 1 | 1 | 1 | 1 | 1 | 0 | 3 | 1 | 19
  Vomiting | 0 | 2 | 1 | 2 | 0 | 2 | 1 | 3 | 15
  Fatigue | 0 | 1 | 1 | 1 | 1 | 2 | 1 | 2 | 18
  Decreased appetite | 1 | 0 | 0 | 1 | 1 | 2 | 1 | 1 | 16
  Anaemia | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 9
  Aspartate aminotransferase increased | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 10
  Dysgeusia | 0 | 1 | 0 | 2 | 2 | 2 | 0 | 2 | 6

7. Secondary Outcome: Number of Participants Reporting a Treatment Emergent Adverse Events With a CTCAE Grade ≥3 During Treatment With PLX3397 (Dose Escalation, Part 1 and Dose Expansion, Part 2)
Description: Data reported are Treatment Emergent Adverse Events with a CTCAE Grade ≥3 During Treatment that are ≥10% Occurrence in all patients.
Time Frame: 1 year post dose
Population: Adverse events were assessed in the Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: 800 mg/Day | Part 1: 1000 mg/Day | Part 1: 1200 mg/Day | Part 1: 1400 mg/Day | Part 1: 2000 mg/Day | Part 1: 3000 mg/Day | Part 1: 4000 mg/Day | Part 1: 5000 mg/Day | Part 2: 3000 mg/Day
Number analyzed (Participants) | 3 | 7 | 3 | 3 | 3 | 6 | 5 | 4 | 56
Participants
  At least 1 AE with CTCAE Grade ≥3 | 3 | 7 | 2 | 3 | 2 | 5 | 5 | 4 | 50
  Febrile neutropenia | 1 | 5 | 1 | 3 | 1 | 1 | 2 | 2 | 22
  Anaemia | 0 | 1 | 0 | 1 | 1 | 0 | 2 | 1 | 9
  Thrombocytopenia | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 3 | 7
  Sepsis | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 10
  Platelet count decreased | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 10
  Fatigue | 2 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 3

8. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Chemistry and Hematology Values Reported as Adverse Events (AE) During Treatment With PLX3397 (Dose Escalation, Part 1 and Dose Expansion, Part 2)
Time Frame: 1 year post dose
Population: Adverse events were assessed in the Safety Population.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1: 4000 mg/Day: Participants with relapsed or refractory acute myeloid leukemia (AML) who received PLX3397 4000 mg/day.
Arm/Group | Part 1: 800 mg/Day | Part 1: 1000 mg/Day | Part 1: 1200 mg/Day | Part 1: 1400 mg/Day | Part 1: 2000 mg/Day | Part 1: 3000 mg/Day | Part 1: 4000 mg/Day | Part 1: 5000 mg/Day | Part 2: 3000 mg/Day
Number analyzed (Participants) | 3 | 7 | 3 | 3 | 3 | 6 | 5 | 4 | 56
Participants
  Anaemia | 0 | 1 | 1 | 1 | 1 | 0 | 2 | 3 | 15
  Hypokalaemia | 1 | 0 | 1 | 2 | 0 | 1 | 2 | 2 | 13
  Aspartate aminotransferase increased | 0 | 1 | 0 | 0 | 2 | 1 | 1 | 1 | 13
  Thrombocytopenia | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 3 | 9
  Hypomagnesmia | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 10
  Hypocalcaemia | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 8
  Platelet count decreased | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 12
  Blood alkaline phosphatase increase | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 10
  Hyperglycaemia | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 9
  Hyponatraemia | 0 | 2 | 0 | 0 | 1 | 2 | 0 | 1 | 5
  Alanine aminotransferase increased | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 6
  Blood bilirubin increased | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 7
  Hypoalbuminaemia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 8
  Hypophosphataemia | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 7
  Transaminases increased | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 5
  White blood cell count decreased | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 7
  Neutropenia | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 4
  Lymphocyte count decreased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7
  Neutrophil count decreased | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 6
  Leukocytosis | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2
  Blood cholesterol increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
  Hyperbilirubinaemia | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Hyperuricaemia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
  Activated partial thromboplastin time prolonged | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Blood urea decreased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Blood uric acid increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  Leukopenia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Hyperchloraemia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Hyperkalaemia | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Bilirubin conjugated increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Blast cell count increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Blood albumin decreased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Blood chloride increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Blood creatinine phosphokinase increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Blood fibrinogen decreased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Carbon monoxide diffusing capacity decreased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Gamma glutamyl transferase increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Globulins increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  INR increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Lipase increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Myeloblast count increased | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Troponin increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  White blood cell count increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Hypernatraemia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Hyperphosphataemia | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

9. Other Pre Specified Outcome: A Summary of Time From Initial Dosing to First and Best Response, Modified Response Criteria in Patient Treated With PLX3397 (Dose Expansion, Part 2)
Time Frame: 1 year post dose
Population: Efficacy analyses were assessed in Part 2 Efficacy Population
Measure: Median (90% Confidence Interval); unit: days
Arm/Group | Part 2: 3000 mg/Day
Number analyzed (Participants) | 11
days
  Time to First Response | 29 [26 to 30]
  Time to Best Response | 30 [26 to 55]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from after the first dose to 30 days after the last dose.
Description: Adverse events that emerge (or worsen) after the first dose of study drug and within 30 days after the last dose.
Arm/Group | Part 1: 800 mg/Day | Part 1: 1000 mg/Day | Part 1: 1200 mg/Day | Part 1: 1400 mg/Day | Part 1: 2000 mg/Day | Part 1: 3000 mg/Day | Part 1: 4000 mg/Day | Part 1: 5000 mg/Day | Part 2: 3000 mg/Day
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/7 | 0/3 | 0/3 | 0/3 | 0/6 | 0/5 | 1/4 | 5/56
Serious Adverse Events (participants affected / at risk) | 1/3 | 5/7 | 2/3 | 1/3 | 2/3 | 5/6 | 4/5 | 4/4 | 39/56
Other Adverse Events (participants affected / at risk) | 3/3 | 7/7 | 3/3 | 3/3 | 3/3 | 6/6 | 5/5 | 4/4 | 56/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: 800 mg/Day (N=3) | Part 1: 1000 mg/Day (N=7) | Part 1: 1200 mg/Day (N=3) | Part 1: 1400 mg/Day (N=3) | Part 1: 2000 mg/Day (N=3) | Part 1: 3000 mg/Day (N=6) | Part 1: 4000 mg/Day (N=5) | Part 1: 5000 mg/Day (N=4) | Part 2: 3000 mg/Day (N=56)
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 9
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 3
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Device related infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 4 | 1 | 0 | 1 | 1 | 2 | 2 | 17
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fungaemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Herpes zoster disseminated (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Streptococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nervous system disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urethral haemorrhage (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Capillary leak syndrome (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malignant hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abscess intestinal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Actinomycosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cerebral toxoplasmosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Enterococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Perirectal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: 800 mg/Day (N=3) | Part 1: 1000 mg/Day (N=7) | Part 1: 1200 mg/Day (N=3) | Part 1: 1400 mg/Day (N=3) | Part 1: 2000 mg/Day (N=3) | Part 1: 3000 mg/Day (N=6) | Part 1: 4000 mg/Day (N=5) | Part 1: 5000 mg/Day (N=4) | Part 2: 3000 mg/Day (N=56)
Diarrhoea (Gastrointestinal disorders) | 3 | 2 | 1 | 2 | 1 | 3 | 4 | 2 | 27
Nausea (Gastrointestinal disorders) | 3 | 1 | 3 | 3 | 0 | 3 | 1 | 3 | 24
Vomiting (Gastrointestinal disorders) | 0 | 3 | 1 | 3 | 0 | 3 | 2 | 3 | 18
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 2 | 0 | 1 | 8
Constipation (Gastrointestinal disorders) | 0 | 2 | 0 | 2 | 0 | 1 | 0 | 0 | 10
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 2
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 4
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Angina bullosa haemorrhagica (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Anorectal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breath odour (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 4
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Gingival hyperplasia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 5
Ileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Large intestinal ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lip ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Proctitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Retching (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Swollen tongue (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Tongue disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tongue ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Fatigue (General disorders) | 3 | 3 | 2 | 2 | 1 | 2 | 1 | 3 | 25
Pyrexia (General disorders) | 2 | 3 | 0 | 0 | 0 | 2 | 1 | 1 | 8
Oedema peripheral (General disorders) | 1 | 2 | 1 | 2 | 0 | 2 | 0 | 0 | 8
Chills (General disorders) | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 2 | 3
Face oedema (General disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 2 | 6
Mucosal dryness (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 4
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Malaise (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Axillary pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Catheter site erythema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Feeling of body temperature change (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypothermia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion site erythema (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infusion site swelling (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Injection site haemorrhage (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nodule (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 4
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Decreased appetite (Metabolism and nutrition disorders) | 1 | 3 | 0 | 2 | 1 | 2 | 2 | 2 | 20
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 3 | 0 | 1 | 2 | 2 | 13
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 8
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 1 | 2 | 0 | 1 | 5
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 10
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 9
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 7
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 8
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1 | 2 | 4 | 2 | 2 | 13
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 3 | 1 | 1 | 2 | 1 | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0 | 1 | 1 | 0 | 1 | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 1 | 0 | 1 | 1 | 0 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 5 | 1 | 3 | 1 | 1 | 2 | 2 | 22
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1 | 1 | 0 | 2 | 3 | 15
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 3 | 9
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 4
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Spleen disorder (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Splenic infarction (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
Pneumonia (Infections and infestations) | 0 | 2 | 0 | 1 | 0 | 1 | 1 | 0 | 6
Candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 10
Clostridial infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Device related infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Streptococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 6
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Enterobacter infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enterococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fungaemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Herpes zoster disseminated (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Mucosal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia klebsiella (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia staphylococcal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin candida (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Urinary tract infection bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 1 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 7
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 3
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Hair colour changes (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 9
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Purpura (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 10
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Facial wasting (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hair disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin tightness (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 2 | 2 | 2 | 0 | 2 | 7
Headache (Nervous system disorders) | 0 | 2 | 1 | 1 | 0 | 1 | 0 | 1 | 6
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 9
Lethargy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 5
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Clumsiness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypersomnia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sensory disturbance (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 7
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Eye swelling (Eye disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blepharitis (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Conjunctival hyperaemia (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eyelid oedema (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Trichiasis (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 2 | 1 | 1 | 1 | 13
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 6
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 10
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 5
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 7
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 4
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 12
Cardiac murmur (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myeloblast count increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 6
Spleen palpable (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Weight increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 7
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 2 | 0 | 0 | 1 | 1 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Soft tissue mass (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 3
Agitation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2
Mental status changes (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 4
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 4
Delirium (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hallucination (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 2 | 8
Hypotension (Vascular disorders) | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 3
Capillary leak syndrome (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Urethral haemorrhage (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hepatic lesion (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatosplenomegaly (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Liver disorder (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Leukaemia cutis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Deafness (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Influenza A (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No